CLINICAL TRIAL: NCT01759784
Title: Safety of Intraventricular Injection of Bone Marrow Derived Mesenchymal Stem Cell in Patients With ALS
Brief Title: Intraventricular Transplantation of Mesenchymal Stem Cell in Patients With ALS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The stereotaxis can be threatful for the patients because of respiratory insufficiency
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Nerve-004
Record Dates: First submitted 2012-12-29; First posted 2013-01-03 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2012-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: mesenchymal stem cell intraventricular injection ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Injections, Intraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell recipient (Experimental): The patients who underwent mesenchymal stem cell transplantation.
  Interventions: Biological: Intraventricular injection

INTERVENTIONS:
Biological: Intraventricular injection — intraventricular injection of mesenchymal stem cell by stereo taxi in patients with ALS
  Other Names: intraventricular injection of mesenchymal stem cell by stereotaxis

SUMMARY:
ALS is a debilitating disease with varied etiology characterized by rapidly progressive weakness, muscle atrophy and fasciculations, muscle spasticity, difficulty speaking (dysarthria), difficulty swallowing (dysphagia), and difficulty breathing (dyspnea). ALS is the most common of the five motor neuron diseases.Riluzole (Rilutek) is the only treatment that has been found to improve survival but only to a modest extent. It lengthens survival by several months, and may have a greater survival benefit for those with a bulbar onset. It also extends the time before a person needs ventilation support.Stem cell transplantation is a new hopeful way to improve the patients conditions and reduce the period of disabilities.

DETAILED DESCRIPTION:
In this study our purpose is to evaluate the safety of intraventricular injection of bone marrow derived mesenchymal stem cell.the patients who are eligible,underwent bone marrow aspiration.after cell separation and preparation,the patients underwent mesenchymal stem cell intraventricular injection by stereotaxis.after injection he will be under observed in ICU to monitor the adverse events(allergic and neurological side effects).patients are followed 1th,3th ,6th and 12 months after injection and each time these parameters are checked:ALS-FRS,EMG-NCV,FVC,side effect check list.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-65
* both gender
* duration of disease<2 years
* FVC>40% ALS-FRS>26

Exclusion Criteria:

* neurological and psychiatric concomitant disease
* concomitant systemic disease
* treatment with corticosteroid,Ig,immunosuppressive during 12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
fever | 48hours
  evaluation the rate of fever 48hours after stem cell injection
unconsciousness | 6months
  evaluation the rate of unconsciousness during 6months after stem cell injection.
brain hematoma | 48hours
  Evaluation the rate of hematoma 48hours after stem cell injection.
vomiting | 48hours
  evaluation the rate of vomiting 48hours after stem cell injection.

SECONDARY OUTCOMES:
ALS-FRS | 6months
  evaluation the improvement of ALS-FRS 6months after stem cell injection.
EMG-NCV | 6months
  evaluation the improvement of EMG-NCV after stem cell injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan department of degenerative medicine,Head of Royan celltherapy center; Ali Reza Zali, MD, Study Director — Head of Neurosurgery research center of Shahid Beheshti University
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org